CLINICAL TRIAL: NCT00084838
Title: A Phase II Study of Intrathecal and Systemic Chemotherapy With Radiation Therapy for Children With Central Nervous System Atypical Teratoid/Rhabdoid Tumor (AT/RT) Tumor
Brief Title: Chemotherapy Combined With Radiation Therapy for Newly Diagnosed CNS AT/RT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Mark W. Kieran, MD, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02-294 DFCI; P30CA006516 (NIH)
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Results first posted 2015-12-24 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-12

CONDITIONS: Central Nervous System Tumor, Pediatric
Keywords: childhood atypical teratoid/rhabdoid tumor
MeSH Terms: conditions — Central Nervous System Neoplasms; Rhabdoid Tumor | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; Cisplatin; Cyclophosphamide; Cytarabine; Dexrazoxane; Razoxane; Doxorubicin; Etoposide; Leucovorin; Methotrexate; Temozolomide; Hydrocortisone; Vincristine; Radiotherapy; Dactinomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Multi-agent Intrathecal and Systemic CT with RT (mod IRS III) (Experimental): Pre-irradiation induction therapy (wks 1-6); Chemoradiation induction therapy (wks 7-12); Post-radiation induction therapy (wks 13-18); Maintenance therapy (wks 19-44); Continuation therapy (wks 45-51)
  Induction Chemotherapy: CT backbone of the IRS-III regimen [vincristine, dactinomycin, cyclophosphamide (specifically, in combination), cisplatin, doxorubicin, and imidazole carboximide (DTIC)] was modified to incl temozolomide in lieu of DTIC. Pts w/ M0 dz (and initially positive CSF cytology) rcvd intrathecal (IT) CT (alt btwn intralumbar and intraventricular routes) w/ methotrexate, cytarabine, and hydrocortisone, coinciding with a cycle of CT.
  Radiation Therapy: Pts w/ M0 dz OR M+ dz aged <3y received focal RT (3D conformal or intensity-modulated delivery). Pts >3y w/ M+ dz rcvd craniospinal irradiation.
  Continuation Therapy: Pts treated with either non-doxorubicin or doxorubicin dose therapy if receiving CSI or mediastinal radiotherapy or not, respectively.
  Interventions: Biological: filgrastim; Drug: cisplatin; Drug: cyclophosphamide; Drug: cytarabine; Drug: dexrazoxane hydrochloride; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: leucovorin calcium; Drug: methotrexate; Drug: temozolomide; Drug: therapeutic hydrocortisone; Drug: vincristine sulfate; Radiation: radiation therapy; Drug: Dactinomycin

INTERVENTIONS:
Biological: filgrastim
  Other Names: filgrastim XM02; G-CSF
Drug: cisplatin
  Other Names: CACP; cis-DDP; cis-diamminedichloro platinum (II); cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cismaplat; Platinol
Drug: cyclophosphamide
  Other Names: Ciclofosfamida; Ciclofosfamide; Claphene; CP monohydrate; CPM; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphanum; Cytophosphane; Mitoxan; Syklofosfamid; Zytoxan; Clafen; Cytoxan; Neosar
Drug: cytarabine
  Other Names: arabinofuranosylcytosine; arabinosylcytosine; aracytidine; beta-cytosine arabinoside; cytarabine hydrochloride; cytarabinum; cytosine arabinoside; cytosine arabinosine hydrochloride; Cytosar-U; Tarabine PFS
Drug: dexrazoxane hydrochloride
  Other Names: Totect; Zinecard
Drug: doxorubicin hydrochloride
  Other Names: Adriamycin PFS; Adriamycin RDF
Drug: etoposide
  Other Names: VP-16
Drug: leucovorin calcium
  Other Names: folinate calcium; folinic acid
Drug: methotrexate
Drug: temozolomide
  Other Names: Temodar, Methazolastone, Temodal, TMZ, CCRG-81045
Drug: therapeutic hydrocortisone
Drug: vincristine sulfate
  Other Names: leurocristine sulfate; Vincasar PFS
Radiation: radiation therapy
Drug: Dactinomycin
  Other Names: ACT-D; actinomycin C1; actinomycin D; actinomycin I1; actinomycin IV; actinomycin X 1; actinomycin-[thr-val-pro-sar-meval]; AD; dactinomycine; meractinomycin

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Giving more than one chemotherapy drug with radiation therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving intrathecal and systemic combination chemotherapy together with radiation therapy works in treating young patients with newly diagnosed central nervous system (CNS) atypical teratoid/rhabdoid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy of intensive systemic and intrathecal chemotherapy and radiotherapy, in terms of medial survival, in children with newly diagnosed central nervous system atypical teratoid/rhabdoid tumors in comparison with historical outcomes from prior trials.

Secondary

* Determine the toxicity profile and tolerability of this regimen in these patients.
* Determine the chemosensitivity of these patients' tumors by Magnetic Resonance Imaging (MRI) after an attempt at maximum surgical resection after 2 courses of this regimen.
* Determine the predictive value of the INI-1 gene mutation in determining prognosis by comparing tumor samples from patients with vs without this mutation treated with this regimen.

STATISTICAL DESIGN: This was a single arm design evaluating median overall survival. The chosen historical control estimate of 7 months was based on 2 large multi-institutional studies in a similar setting and the alternative of 20.5 months based on a DFCI pilot study. There was 90% power to detect this improvement assuming 1-sided 0.10 alpha and 17 eligible patients. Sample size (n=20 patients) was inflated for expected 10-15% ineligible rate.

TREATMENT: Induction chemotherapy was required to be initiated within 50 days of the most definitive surgery.

* Central Nervous System (CNS)/intrathecal therapy: All patients with M0 disease receive triple intrathecal (IT) chemotherapy comprising methotrexate (MTX), cytarabine, and hydrocortisone on day 1 of weeks 1, 2, 4, 7, 13, 19, 27, 33, 39, 45, and 51 followed by oral or intravenous (IV) leucovorin calcium given 24 hours after each MTX dose. Patients with initially positive cerebrospinal fluid (CSF) cytology (M+) receive triple IT chemotherapy weekly until 2 consecutive CSF samples are negative for malignant cells.
* Pre-irradiation induction therapy (weeks 1-6): Patients receive vincristine IV on day 1 of weeks 1-6; cisplatin IV over 8 hours on day 1 and doxorubicin IV continuously over 48 hours beginning on day 2 of weeks 1 and 4; cyclophosphamide IV continuously over 72 hours beginning on day 2 of week 1; etoposide IV over 1 hour on days 1-3 of week 4; and filgrastim (G-CSF) subcutaneously (SC) beginning on day 6 of week 1 and day 4 of week 4 and continuing until blood counts recover.
* Induction chemoradiotherapy (weeks 7-12): Patients receive vincristine IV on day 1 of weeks 7-12; cisplatin IV over 8 hours on day 1, cyclophosphamide IV over 1 hour on day 2, etoposide IV over 1 hour on days 1-3 of weeks 7 and 10; and granulocyte-colony stimulating factor (G-CSF) subcutaneous (SC) daily beginning on day 4 of weeks 7 and 10 and continuing until blood counts recover. Patients with M0 disease and patients under 3 years of age with M+ disease undergo radiotherapy to the primary tumor daily on weeks 7-12. Patients 3 years of age and over with M+ disease undergo craniospinal irradiation (CSI) daily on weeks 7-12 until negative cerebral spinal fluid (CSF) cytology is achieved.
* Post-radiation induction therapy (weeks 13-18): Patients receive vincristine IV on day 1 of weeks 13 and 16; doxorubicin and cyclophosphamide as in pre-irradiation induction therapy beginning on day 1 of week 13; cyclophosphamide IV over 1 hour on days 1-3 of week 16; dactinomycin IV on days 1-5 of week 16; and G-CSF SC daily beginning on day 6 of weeks 13 and 16 and continuing until blood counts recover.
* Maintenance chemotherapy (weeks 19-42): Patients receive vincristine IV on day 1 of weeks 27, 33, and 39 and days 1 and 5 of weeks 30, 36, and 42; doxorubicin and cyclophosphamide as in pre-irradiation induction beginning on day 1 of weeks 27 and 33; doxorubicin IV over 15 minutes and dexrazoxane (DX) IV over 15 minutes on days 1 and 2 of week 39; cyclophosphamide IV over 1 hour on days 1-3 of weeks 30, 36, 39, and 42; dactinomycin IV on days 1-5 of weeks 30, 36, and 42 and on day 1 of weeks 19 and 23; oral temozolomide on days 1-5 of weeks 19 and 23; and G-CSF SC daily beginning on day 6 of weeks 19, 23, 30, 36, and 42, day 5 of weeks 27 and 33, and day 4 of week 39 and continuing until blood counts recover.
* Doxorubicin continuation therapy (for patients not receiving CSI and mediastinal radiotherapy)(weeks 45-51): Patients receive vincristine IV on day 1 of weeks 45, 48, and 51 and day 5 of week 48; doxorubicin IV over 15 minutes and DX IV over 15 minutes on days 1 and 2 of weeks 45 and 51; cyclophosphamide IV over 1 hour on days 1-3 of weeks 45, 48, and 51; dactinomycin IV on days 1-5 of week 48; and G-CSF SC daily beginning on day 4 of weeks 45 and 51 and day 6 of week 48 and continuing until blood counts recover.
* Non-doxorubicin continuation therapy (for patients receiving CSI or mediastinal radiotherapy)(weeks 45-51): Patients receive cyclophosphamide and G-CSF as in doxorubicin continuation therapy; vincristine IV on days 1 and 5 of weeks 45, 48, and 51; and dactinomycin IV on days 1-5 of weeks 45, 48, and 51.

Treatment continues in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary intracranial Central Nervous System (CNS) atypical teratoid/rhabdoid tumor OR
* Tumor tissue that possesses the INI-1 gene mutation
* No metastases that disseminate outside the CNS by abdominal and chest computer tomography (CT) scans, kidney imaging, and bone marrow biopsy

  * No obstruction of cerebrospinal fluid (CSF) flow by CSF flow study
* Definitive surgical resection of tumor within the past 35 days

PATIENT CHARACTERISTICS:

Age

* 18 and under

Performance status

* Karnofsky 50-100% OR
* Lansky 50-100%

Life expectancy

* Not specified

Hematopoietic

* Hemoglobin > 10 g/dL
* Absolute neutrophil count > 1,000/mm^3
* Platelet count > 100,000/mm^3

Hepatic

* Bilirubin ≤ 1.5 mg/dL
* SGPT < 10 times normal

Renal

* Creatinine ≤ 1.5 times normal

Other

* Willing to have placement of central venous access line

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy

Endocrine therapy

* Prior steroids allowed

Radiotherapy

* No prior radiotherapy

Surgery

* See Disease Characteristics

Other

* No other prior or concurrent investigational agents
* Concurrent anticonvulsant agents allowed

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2003-02; Primary Completion 2008-02 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark W. Kieran, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (12):
- United States (12):
  - Stanford Cancer Center, Stanford, California
  - Yale Cancer Center, New Haven, Connecticut
  - AFLAC Cancer Center and Blood Disorders Service of Children's Healthcare of Atlanta - Scottish Rite Campus, Atlanta, Georgia
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Children's Hospital Boston, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas

REFERENCES:
- [Result] Chi SN, Zimmerman MA, Yao X, Cohen KJ, Burger P, Biegel JA, Rorke-Adams LB, Fisher MJ, Janss A, Mazewski C, Goldman S, Manley PE, Bowers DC, Bendel A, Rubin J, Turner CD, Marcus KJ, Goumnerova L, Ullrich NJ, Kieran MW. Intensive multimodality treatment for children with newly diagnosed CNS atypical teratoid rhabdoid tumor. J Clin Oncol. 2009 Jan 20;27(3):385-9. doi: 10.1200/JCO.2008.18.7724. Epub 2008 Dec 8. PMID 19064966

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment Sep 2004 to Sep 2006 at 9 institutions.
Groups:
- Multi-agent Intrathecal and Systemic CT With RT (Modified IRS: Pre-irradiation induction therapy (wks 1-6); Chemoradiation induction therapy (wks 7-12); Post-radiation induction therapy (wks 13-18); Maintenance therapy (wks 19-44); Continuation therapy (wks 45-51) Induction Chemotherapy: CT backbone of the IRS-III regimen [vincristine, dactinomycin, cyclophosphamide (specifically, in combination), cisplatin, doxorubicin, and imidazole carboximide (DTIC)] was modified to incl temozolomide in lieu of DTIC. Pts w/ M0 dz (and initially positive CSF cytology) rcvd intrathecal (IT) CT (alt btwn intralumbar and intraventricular routes) w/ methotrexate, cytarabine, and hydrocortisone, coinciding with a cycle of CT.
  Radiation Therapy: Pts w/ M0 dz OR M+ dz aged <3y received focal RT (3D conformal or intensity-modulated delivery). Pts >3y w/ M+ dz rcvd craniospinal irradiation.
  Continuation Therapy: Pts treated with either non-doxorubicin or doxorubicin dose therapy if receiving CSI or mediastinal radiotherapy or not, respectively.
Period: Overall Study
Arm/Group | Multi-agent Intrathecal and Systemic CT With RT (Modified IRS
Started | 25
Eligible and Treated | 20 (4 ineligible pts upon central path review (n=3) and per DFCI IRB (n=1); 1 pt withdrew before rcv trt)
Completed | 12
Not Completed | 13
Not completed — Death | 1
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 1
Not completed — Progressive Disease | 4
Not completed — Pt Non-Compliance | 1
Not completed — Ineligible | 4

BASELINE CHARACTERISTICS:
Groups:
- Multi-agent Intrathecal & Systemic CT w/ RT (Modified IRS III): Pre-irradiation induction therapy (wks 1-6); Chemoradiation induction therapy (wks 7-12); Post-radiation induction therapy (wks 13-18); Maintenance therapy (wks 19-44); Continuation therapy (wks 45-51) Induction Chemotherapy: CT backbone of the IRS-III regimen [vincristine, dactinomycin, cyclophosphamide (specifically, in combination), cisplatin, doxorubicin, and imidazole carboximide (DTIC)] was modified to incl temozolomide in lieu of DTIC. Pts w/ M0 dz (and initially positive CSF cytology) rcvd intrathecal (IT) CT (alt btwn intralumbar and intraventricular routes) w/ methotrexate, cytarabine,and hydrocortisone, coinciding with a cycle of CT.
  Radiation Therapy: Pts w/ M0 dz OR M+ dz aged <3y received focal RT (3D conformal or intensity-modulated delivery). Pts >3y w/ M+ dz rcvd craniospinal irradiation.
  Continuation Therapy: Pts treated with either non-doxorubicin or doxorubicin dose therapy if receiving CSI or mediastinal radiotherapy or not, respectively.
Arm/Group | Multi-agent Intrathecal & Systemic CT w/ RT (Modified IRS III)
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: years] | 2.2 [0.2 to 19]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 20
Chang Stage [Number; unit: participants] — Chang staging: M0 is non-metastatic disease. M1 is CSF +ve disease which means that the tumor cells are found floating in the spinal fluid, M2 is localized metastatic disease and M3 is disseminated bulk disease.
  participants
    M0 | 14
    M2 | 1
    M3 | 5

OUTCOME MEASURES:

1. Primary Outcome: 2-yr Overall Survival
Description: Overall survival is defined as the time from date of diagnosis to death or date of last follow-up. 2-year overall survival is the probability of patients remaining alive at 2-years from study entry estimated using Kaplan-Meier (KM) methods which censors patients at date of last follow-up. Precision of this conditional probability estimate was measured in terms of standard error. Median OS, the original primary endpoint, was not estimable based on the Kaplan-Meier method because of insufficient follow-up.
Time Frame: Patients are followed for survival up to 5 yrs post-therapy completion or death; As of this analysis, median follow-up among survivors was 31 months with the longest follow-up being 40 months.
Population: The analysis dataset is comprised of all eligible and treated patients.
Measure: Number; unit: probability
Arm/Group | Multi-agent Intrathecal and Systemic CT With RT (Modified IRS
Number analyzed (Participants) | 20
probability | 0.70

2. Secondary Outcome: Pre-Radiation Therapy Chemotherapeutic Response
Description: Response pre-RT/post-CT was defined as follows with overall response defined as achieving PR or CR.
  Complete Response (CR): Complete resolution of all initially demonstrable tumor on MRI or CT evaluation w/o appearance of any new areas of disease; negative CSF cytology. Partial Response (PR): >/= 50% decrease in the sum of the products of the maximum perpendicular diameters of the tumor (sum LD) relative to baseline w/o appearance of any new areas of disease; CSF cytology unchanged from that at diagnosis or clearing after being initially positive Stable Disease (SD): <50% decrease in the sum LD w/o appearance of any new areas of disease; CSF cytology unchanged from that at diagnosis or clearing after being initially positive Progressive Disease (PD): >/= 25% increase in the sum LD relative to baseline, or the appearance of any new areas of disease or appearance of positive cytology after two consecutive negative samples.
Time Frame: Assessed at study entry and pre-RT/post-CT at week 7.
Population: The pre-RT CT response evaluable population is defined as patients who completed chemotherapy per protocol.
Measure: Number (90% Confidence Interval); unit: proportion of evaluable patients
Arm/Group | Multi-agent Intrathecal and Systemic CT With RT (Modified IRS
Number analyzed (Participants) | 12
proportion of evaluable patients | 0.58 [0.32 to 0.82]

3. Other Pre Specified Outcome: Grade 3/4 Events
Description: All Grade 3-4 events based on CTCAEv2 as reported on case report forms.
Time Frame: Assessed during therapy up to 30 days post-therapy completion which is approximately 55 weeks for patients who completed therapy.
Population: The analysis population excludes 1 patient who withdrew before treatment.
Measure: Number; unit: adverse events
Arm/Group | Multi-agent Intrathecal and Systemic CT With RT (Mod IRS III)
Number analyzed (Participants) | 24
adverse events | 1021

4. Other Pre Specified Outcome: Grade 3-4 Auditory/Hearing Events
Description: All Grade 3-4 Auditory/Hearing events based on CTCAEv2 as reported on case report forms.
Time Frame: as for outcome 3
Population: The analysis population excludes 1 patient who withdrew before treatment.
Measure: Number; unit: adverse events
Groups:
- Multi-agent Intrathecal and Systemic CT With RT (Mod IRS III): Pre-irradiation induction therapy (wks 1-6); Chemoradiation induction therapy (wks 7-12); Post-radiation induction therapy (wks 13-18); Maintenance therapy (wks 19-44); Continuation therapy (wks 45-51)
  Induction Chemotherapy: CT backbone of the IRS-III regimen [vincristine, dactinomycin, cyclophosphamide (specifically, in combination), cisplatin, doxorubicin, and imidazole carboximide (DTIC)] was modified to incl temozolomide in lieu of DTIC. Pts w/ M0 dz (and initially positive CSF cytology) rcvd intrathecal (IT) CT (alt btwn intralumbar and intraventricular routes) w/ methotrexate, cytarabine, and hydrocortisone, coinciding with a cycle of CT.
  Radiation Therapy: Pts w/ M0 dz OR M+ dz aged <3y received focal RT (3D conformal or intensity-modulated delivery). Pts >3y w/ M+ dz rcvd craniospinal irradiation.
  Continuation Therapy: Pts treated with either non-doxorubicin or doxorubicin dose therapy if receiving CSI or mediastinal radiotherapy or not, respectively.
  filgrastim
Arm/Group | Multi-agent Intrathecal and Systemic CT With RT (Mod IRS III)
Number analyzed (Participants) | 24
adverse events | 8

5. Other Pre Specified Outcome: Grade 3-4 Blood/Bone Marrow Events
Description: All Grade 3-4 Blood/Bone Marrow events based on CTCAEv2 as reported on case report forms.
  Arm Name
Time Frame: as for outcome 3
Population: The analysis population excludes 1 patient who withdrew before treatment.
Measure: Number; unit: adverse events
Arm/Group | Multi-agent Intrathecal and Systemic CT With RT (Mod IRS III)
Number analyzed (Participants) | 24
adverse events | 564

6. Other Pre Specified Outcome: Grade 3-4 Gastrointestinal Events
Description: All Grade 3-4 Gastrointestinal events based on CTCAEv2 as reported on case report forms.
Time Frame: as for outcome 3
Population: The analysis population excludes 1 patient who withdrew before treatment.
Measure: Number; unit: adverse events
Arm/Group | Multi-agent Intrathecal and Systemic CT With RT (Mod IRS III)
Number analyzed (Participants) | 24
adverse events | 139

7. Other Pre Specified Outcome: Grade 3-4 Metabolic/Laboratory Events
Description: All Grade 3-4 Metabolic/Laboratory events based on CTCAEv2 as reported on case report forms.
Time Frame: as for outcome 3
Population: The analysis population excludes 1 patient who withdrew before treatment.
Measure: Number; unit: adverse events
Arm/Group | Multi-agent Intrathecal and Systemic CT With RT (Mod IRS III)
Number analyzed (Participants) | 24
adverse events | 128

8. Other Pre Specified Outcome: Grade 3-4 Infection/Febrile Neutropenia Events
Description: All Grade 3-4 Infection/Febrile Neutropenia events based on CTCAEv2 as reported on case report forms.
Time Frame: as for outcome 3
Population: The analysis population excludes 1 patient who withdrew before treatment.
Measure: Number; unit: adverse events
Arm/Group | Multi-agent Intrathecal and Systemic CT With RT (Mod IRS III)
Number analyzed (Participants) | 24
adverse events | 49

9. Other Pre Specified Outcome: Grade 3-4 Neurology Events
Description: All Grade 3-4 Neurology events based on CTCAEv2 as reported on case report forms.
Time Frame: as for outcome 3
Population: The analysis population excludes 1 patient who withdrew before treatment.
Measure: Number; unit: adverse events
Arm/Group | Multi-agent Intrathecal and Systemic CT With RT (Mod IRS III)
Number analyzed (Participants) | 24
adverse events | 45

10. Other Pre Specified Outcome: Grade 3-4 Pain Events
Description: All Grade 3-4 Pain events based on CTCAEv2 as reported on case report forms.
Time Frame: as for outcome 3
Population: The analysis population excludes 1 patient who withdrew before treatment.
Measure: Number; unit: adverse events
Arm/Group | Multi-agent Intrathecal and Systemic CT With RT (Mod IRS III)
Number analyzed (Participants) | 24
adverse events | 31

11. Other Pre Specified Outcome: Grade 3-4 Constitutional Events
Description: All Grade 3-4 Constitutional events based on CTCAEv2 as reported on case report forms.
Time Frame: as for outcome 3
Population: The analysis population excludes 1 patient who withdrew before treatment.
Measure: Number; unit: adverse events
Arm/Group | Multi-agent Intrathecal and Systemic CT With RT (Mod IRS III)
Number analyzed (Participants) | 24
adverse events | 22

12. Other Pre Specified Outcome: Grade 3-4 Muscloskeletal Events
Description: All Grade 3-4 Muscloskeletal events based on CTCAEv2 as reported on case report forms.
Time Frame: as for outcome 3
Population: The analysis population excludes 1 patient who withdrew before treatment.
Measure: Number; unit: adverse events
Arm/Group | Multi-agent Intrathecal and Systemic CT With RT (Mod IRS III)
Number analyzed (Participants) | 24
adverse events | 8

13. Other Pre Specified Outcome: Grade 3-4 Hepatic Events
Description: All Grade 3-4 Hepatic events based on CTCAEv2 as reported on case report forms.
Time Frame: as for outcome 3
Population: The analysis population excludes 1 patient who withdrew before treatment.
Measure: Number; unit: adverse events
Arm/Group | Multi-agent Intrathecal and Systemic CT With RT (Mod IRS III)
Number analyzed (Participants) | 24
adverse events | 8

14. Other Pre Specified Outcome: Grade 3-4 Cardiovascular Events
Description: All Grade 3-4 Cardiovascular events based on CTCAEv2 as reported on case report forms.
Time Frame: as for outcome 3
Population: The analysis population excludes 1 patient who withdrew before treatment.
Measure: Number; unit: adverse events
Arm/Group | Multi-agent Intrathecal and Systemic CT With RT (Mod IRS III)
Number analyzed (Participants) | 24
adverse events | 6

15. Other Pre Specified Outcome: Grade 3-4 Pulmonary Events
Description: All Grade 3-4 Pulmonary events based on CTCAEv2 as reported on case report forms.
Time Frame: as for outcome 3
Population: The analysis population excludes 1 patient who withdrew before treatment.
Measure: Number; unit: adverse events
Arm/Group | Multi-agent Intrathecal and Systemic CT With RT (Mod IRS III)
Number analyzed (Participants) | 24
adverse events | 4

16. Other Pre Specified Outcome: Grade 3-4 Renal/Genitourinary Events
Description: All Grade 3-4 Renal/Genitourinary events based on CTCAEv2 as reported on case report forms.
Time Frame: as for outcome 3
Population: The analysis population excludes 1 patient who withdrew before treatment.
Measure: Number; unit: adverse events
Arm/Group | Multi-agent Intrathecal and Systemic CT With RT (Mod IRS III)
Number analyzed (Participants) | 24
adverse events | 4

17. Other Pre Specified Outcome: Grade 3-4 Dermatology Events
Description: All Grade 3-4 Dermatology events based on CTCAEv2 as reported on case report forms.
Time Frame: as for outcome 3
Population: The analysis population excludes 1 patient who withdrew before treatment.
Measure: Number; unit: adverse events
Arm/Group | Multi-agent Intrathecal and Systemic CT With RT (Mod IRS III)
Number analyzed (Participants) | 24
adverse events | 3

18. Other Pre Specified Outcome: Grade 3-4 Hemorrhage Events
Description: All Grade 3-4 Hemorrhage events based on CTCAEv2 as reported on case report forms.
Time Frame: as for outcome 3
Population: The analysis population excludes 1 patient who withdrew before treatment.
Measure: Number; unit: adverse events
Arm/Group | Multi-agent Intrathecal and Systemic CT With RT (Mod IRS III)
Number analyzed (Participants) | 24
adverse events | 1

19. Other Pre Specified Outcome: Grade 3-4 Allergy/Immunology
Description: All Grade 3-4 Allergy/Immunology events based on CTCAEv2 as reported on case report forms.
Time Frame: as for outcome 3
Population: The analysis population excludes 1 patient who withdrew before treatment.
Measure: Number; unit: adverse events
Arm/Group | Multi-agent Intrathecal and Systemic CT With RT (Mod IRS III)
Number analyzed (Participants) | 24
adverse events | 1

ADVERSE EVENTS:
Time Frame: Assessed during therapy up to 30 days post-therapy completion which is approximately 55 weeks for patients who completed therapy.
Description: SAEs were grade 3+ unexpected, treatment-related events deemed notable by the study chair. Accessible adverse event data represents a count of events by toxicity type rather than worst-grade by toxicity type and therefore cannot be reported in the established framework (Affected/At Risk). See secondary outcomes for events by system organ class.
Arm/Group | Multi-agent Intrathecal & Systemic CT w/ RT (Modified IRS III)
Serious Adverse Events (participants affected / at risk) | 4/20
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Multi-agent Intrathecal & Systemic CT w/ RT (Modified IRS III) (N=20)
Sepsis (Infections and infestations) | 1 (1) — Patient died of pneumococcal sepsis
Radiation recall (Nervous system disorders) | 2 (2)
Transverse Myeolitis (Nervous system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
None. Trial was completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less